CLINICAL TRIAL: NCT02069509
Title: Patient Registry of the European Friedreich's Ataxia Consortium for Translational Studies (EFACTS)
Acronym: EFACTS
Status: Completed | Type: Observational
Sponsor: European Friedreich's Ataxia Consortium for Translational Studies (Other)
Responsible Party: Sponsor
Other Study IDs: HEALTH-F2-2010- 242193
Record Dates: First submitted 2014-02-19; First posted 2014-02-24 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Friedreich's Ataxia
Keywords: Friedreich's Ataxia; EFACTS; FRDA
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Biospecimen Retention: Samples With DNA — whole blood, urine, centrifugate of serum, EDTA, citrate blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control research participants: Controls may be family members or recruited elsewhere, heterozygous GAA expansion carriers are allowed
- FRDA patients: with genetically confirmed diagnosis of FRDA

SUMMARY:
This is a multi-centre, multi-national, prospective, observational study of Friedreich's Ataxia (FRDA) with a control group to:

* obtain natural history data on individuals affected by FRDA
* relate clinical assessments and results from proteomic analyses
* expedite identification and recruitment of participants for clinical trials
* develop and validate sensitive and reliable outcome measures for detecting onset and change over the natural course of FRDA which may also be potential outcome measures for use in future clinical trials and clinical care
* plan for future research studies

DETAILED DESCRIPTION:
The EFACTS patient registry integrates prospectively and systematically collected clinical research data (e.g. clinical tests, demographical characteristics) with access to biological specimens (e.g. blood, urine) obtained from individuals with genetically confirmed FRDA and unrelated control research participants.

The EFACTS patient registry started out as a 4-year study and is currently running without a set end date. Eligible subjects are assessed at annual study visits on the clinical symptoms and signs of the disease. At each study visit, general clinical, motor function, cognitive, and Quality of Life assessments are administered. In addition, participants are providing bio samples for the purposes of genetic testing and for research to identify valuable biomarkers of FRDA. Biological specimens and clinical data are made available to qualified scientists within the EFACTS network whose projects are reviewed and approved by the EFACTS Steering Committee. Research projects should aim to advance scientific knowledge towards establishing clinically effective treatments that delay onset and/or slow the progression of the disease.

The EFACTS study will now be converted to a globally harmonized version of the protocol. Data from Europe will continue to be stored in a European database maintained by FARA Europe. While this is a continuation of the study for current patients, the project will be given the new study title UNIFAI to reflect the inclusion of new global sites.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of FRDA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a genetically confirmed diagnosis of FRDA and control research participants.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Disease progression as assessed by clinical examination | Participants are followed with annual assessments

OTHER OUTCOMES:
Transition to UNIFAI | 2010-2024
  The EFACTS study will now be converted to a globally harmonized version of the protocol. Data from Europe will continue to be stored in a European database maintained by FARA Europe. While this is a continuation of the study for current patients, the project will be given the new study title UNIFAI to reflect the inclusion of new global sites.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg B. Schulz, MD, Principal Investigator — University Hospital Aachen, Dept. of Neurology; Paola Giunti, MD, Principal Investigator — University College of London, Institute of Neurology; Caterina Mariotti, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta; Francisco J. Rodriguez de Rivera Garrido, MD, Principal Investigator — La Paz University Hospital, Dept. of Neurology; Alexandra Durr, MD, Principal Investigator — Hôpital Pitié Salpêtrière, ICM; Thomas Klopstock, MD, Principal Investigator — University of Munich, Dept. of Neurology with Friedrich-Baur-Institute; Sylvia Boesch, MD, Principal Investigator — Medical University Innsbruck, Department of Neurology; Gilles Naeije, MD, Principal Investigator — Université Libre de Bruxelles and Cliniques Universitaires de Bruxelles-Hôpital Erasme; Ludger Schöls, MD, Principal Investigator — University of Tübingen, Dept. of Neurology with Hertie-Institute for Clinical Brain Research; Thomas Klockgether, MD, Principal Investigator — University Hospital Bonn, Dept. of Neurology; Georgios Koutsis, MD, Principal Investigator — National and Kapodistrian University of Athens, Neurogenetics Unit; Sinead Murphy, MD, Principal Investigator — Tallaght University Hospital, Department of Neurology; Richard Walsh, MD, Principal Investigator — Tallaght University Hospital, Department of Neurology; Enrico Bertini, MD, Principal Investigator — Bambino Gesù Children's Hospital, Department of Neurosciences; Francesc Palau Martinez, MD, Principal Investigator — Hospital Sant Joan de Déu, Servicio de Neurología; Martin Vyhnálek, MD, Principal Investigator — Motol University Hospital, Centre for Hereditary Ataxias; Mathieu Anheim, MD, Principal Investigator — Hôpital de Hautepierre, Service de Neurologie; Bart van de Warrenburg, MD, Principal Investigator — STICHTING RADBOUD UNIVERSITAIR MEDISCH CENTRUM; Kathrin Reetz, MD, Principal Investigator — University Hospital Aachen, Dept. of Neurology
Locations (16):
- Medical University Innsbruck, Department of Neurology, Innsbruck, Austria
- Université Libre de Bruxelles, Hôpital Erasme, Dpt of Neurology, Brussels, Belgium
- Motol University Hospital, Centre for Hereditary Ataxias, Prague, Czechia
- France (2):
  - Hôpital Pitié Salpêtrière, Bâtiment ICM, Paris
  - Hôpital de Hautepierre, Service de Neurologie, Strasbourg
- Germany (4):
  - University Hospital Aachen, Dept. of Neurology, Aachen
  - University Hospital Bonn, Dept. of Neurology, Bonn
  - University of Munich, Dept. of Neurology, Friedrich-Baur-Institut, Munich
  - University of Tübingen, Dept. of Neurodegenerative Diseases, Hertie-Institute for Clinical Brain Research, Tübingen
- National and Kapodistrian University of Athens, Neurogenetics Unit, Athens, Greece
- Tallaght University Hospital, Department of Neurology, Dublin, Ireland
- Italy (2):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Bambino Gesù Children's Hospital, Department of Neurosciences, Roma
- Spain (2):
  - Hospital Sant Joan de Déu, Servicio de Neurología, Barcelona
  - Hospital Universitario La Paz, Servicio de Neurologia, Madrid
- University College of London, Ataxia Centre, National Hospital for Neurology and Neurosurgery, London, United Kingdom

REFERENCES:
- [Background] Reetz K, Dogan I, Costa AS, Dafotakis M, Fedosov K, Giunti P, Parkinson MH, Sweeney MG, Mariotti C, Panzeri M, Nanetti L, Arpa J, Sanz-Gallego I, Durr A, Charles P, Boesch S, Nachbauer W, Klopstock T, Karin I, Depondt C, vom Hagen JM, Schols L, Giordano IA, Klockgether T, Burk K, Pandolfo M, Schulz JB. Biological and clinical characteristics of the European Friedreich's Ataxia Consortium for Translational Studies (EFACTS) cohort: a cross-sectional analysis of baseline data. Lancet Neurol. 2015 Feb;14(2):174-82. doi: 10.1016/S1474-4422(14)70321-7. Epub 2015 Jan 5. PMID 25566998
- [Derived] Buchholz M, Pfaff M, Iskandar A, Reetz K, Schulz JB, Grobe-Einsler M, Klockgether T, Michalowsky B; EFACTS Study Group. Health-Related Quality of Life in Patients with Friedreich Ataxia Using Mobility Assistive Technologies: Limited Fit of the EQ-5D-3L Mobility Dimension. Neurol Ther. 2025 Feb;14(1):379-398. doi: 10.1007/s40120-024-00694-7. Epub 2024 Dec 30. PMID 39738982
- [Derived] Indelicato E, Reetz K, Maier S, Nachbauer W, Amprosi M, Giunti P, Mariotti C, Durr A, de Rivera Garrido FJR, Klopstock T, Schols L, Klockgether T, Burk K, Pandolfo M, Didszun C, Grobe-Einsler M, Nanetti L, Nenning L, Kiechl S, Dichtl W, Ulmer H, Schulz JB, Boesch S; European Friedreich's Ataxia Consortium for Translational Studies (EFACTS). Predictors of Survival in Friedreich's Ataxia: A Prospective Cohort Study. Mov Disord. 2024 Mar;39(3):510-518. doi: 10.1002/mds.29687. Epub 2023 Dec 23. PMID 38140802
- [Derived] Reetz K, Dogan I, Hilgers RD, Giunti P, Parkinson MH, Mariotti C, Nanetti L, Durr A, Ewenczyk C, Boesch S, Nachbauer W, Klopstock T, Stendel C, Rodriguez de Rivera Garrido FJ, Rummey C, Schols L, Hayer SN, Klockgether T, Giordano I, Didszun C, Rai M, Pandolfo M, Schulz JB; EFACTS study group. Progression characteristics of the European Friedreich's Ataxia Consortium for Translational Studies (EFACTS): a 4-year cohort study. Lancet Neurol. 2021 May;20(5):362-372. doi: 10.1016/S1474-4422(21)00027-2. Epub 2021 Mar 23. PMID 33770527
- [Derived] Indelicato E, Nachbauer W, Eigentler A, Amprosi M, Matteucci Gothe R, Giunti P, Mariotti C, Arpa J, Durr A, Klopstock T, Schols L, Giordano I, Burk K, Pandolfo M, Didszdun C, Schulz JB, Boesch S; EFACTS (European Friedreich's Ataxia Consortium for Translational Studies). Onset features and time to diagnosis in Friedreich's Ataxia. Orphanet J Rare Dis. 2020 Aug 3;15(1):198. doi: 10.1186/s13023-020-01475-9. PMID 32746884
- [Derived] Bonnechere B, Jansen B, Haack I, Omelina L, Feipel V, Van Sint Jan S, Pandolfo M. Automated functional upper limb evaluation of patients with Friedreich ataxia using serious games rehabilitation exercises. J Neuroeng Rehabil. 2018 Oct 4;15(1):87. doi: 10.1186/s12984-018-0430-7. PMID 30286776
- [Derived] Reetz K, Dogan I, Hohenfeld C, Didszun C, Giunti P, Mariotti C, Durr A, Boesch S, Klopstock T, Rodriguez de Rivera Garrido FJ, Schols L, Giordano I, Burk K, Pandolfo M, Schulz JB; EFACTS Study Group. Nonataxia symptoms in Friedreich Ataxia: Report from the Registry of the European Friedreich's Ataxia Consortium for Translational Studies (EFACTS). Neurology. 2018 Sep 4;91(10):e917-e930. doi: 10.1212/WNL.0000000000006121. Epub 2018 Aug 10. PMID 30097477
- [Derived] Tanguy Melac A, Mariotti C, Filipovic Pierucci A, Giunti P, Arpa J, Boesch S, Klopstock T, Muller Vom Hagen J, Klockgether T, Burk K, Schulz JB, Reetz K, Pandolfo M, Durr A, Tezenas du Montcel S; EFACTS group. Friedreich and dominant ataxias: quantitative differences in cerebellar dysfunction measurements. J Neurol Neurosurg Psychiatry. 2018 Jun;89(6):559-565. doi: 10.1136/jnnp-2017-316964. Epub 2017 Dec 26. PMID 29279305
- [Derived] Lad M, Parkinson MH, Rai M, Pandolfo M, Bogdanova-Mihaylova P, Walsh RA, Murphy S, Emmanuel A, Panicker J, Giunti P. Urinary, bowel and sexual symptoms in a cohort of patients with Friedreich's ataxia. Orphanet J Rare Dis. 2017 Sep 26;12(1):158. doi: 10.1186/s13023-017-0709-y. PMID 28950889
- [Derived] Reetz K, Dogan I, Hilgers RD, Giunti P, Mariotti C, Durr A, Boesch S, Klopstock T, de Rivera FJR, Schols L, Klockgether T, Burk K, Rai M, Pandolfo M, Schulz JB; EFACTS Study Group. Progression characteristics of the European Friedreich's Ataxia Consortium for Translational Studies (EFACTS): a 2 year cohort study. Lancet Neurol. 2016 Dec;15(13):1346-1354. doi: 10.1016/S1474-4422(16)30287-3. PMID 27839651
- See also: EFACTS Registry — http://www.e-facts.eu